CLINICAL TRIAL: NCT06082024
Title: The Second Affiliated Hospital of Nanchang University
Brief Title: Correlation Between Perioperative EEG Features and Delirium After General Anesthesia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fuzhou Hua (Other)
Responsible Party: Sponsor-Investigator, Fuzhou Hua, Director, Second Affiliated Hospital of Nanchang University
Organization: Second Affiliated Hospital of Nanchang University (Other)
Other Study IDs: 2023-EEG-1
Record Dates: First submitted 2023-09-05; First posted 2023-10-13 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Perioperative Period; Anesthetic; Postoperative Cognitive Dysfunction; Postoperative Delirium
Keywords: Perioperative period; Anesthetics; Postoperative Cognitive Dysfunction; postoperative delirium
MeSH Terms: conditions — Postoperative Cognitive Complications; Emergence Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- delirium: Patients present with delirium within 7 days after general anesthesia
- non delirium: The patient did not develop delirium for 7 days after general anesthesia

SUMMARY:
The goal of this observational study is to compare the perioperative EEG characteristics and the incidence of short-term cognitive dysfunction in patients with postoperative delirium and non-postoperative delirium after elderly (> 65 years old) patients undergoing major gastrointestinal surgery under general anesthesia. The main question it aims to answer are: • The correlation between postoperative cognitive dysfunction and postoperative EEG features was evaluated.• To analyze the correlation between EEG characteristics and clinical risk factors of delirium after major abdominal gastrointestinal surgery under general anesthesia in elderly patients.Participants will collect EEG before and after operation and collect the incidence of postoperative cognitive function to explore the mechanism of postoperative delirium and predict postoperative cognitive dysfunction.

ELIGIBILITY:
Inclusion Criteria:

1. Education level in primary school or above;
2. Age ≥65 years old, gender is not limited;
3. Good communication ability, language expression ability, mental state and consciousness state;
4. Preoperative simple mental state scale score ≥27 points;
5. no history of craniocerebral diseases;
6. For patients who plan to choose abdominal surgery under general anesthesia, the operation time is expected to be about 2h-4h;
7. ASA anesthesia grade I ~ III;
8. No general anesthesia contraindications;
9. Sign informed consent voluntarily;

Exclusion Criteria:

1. Relative contraindications of general anesthesia: patients with serious heart and lung function diseases, drug allergy history, etc.
2. Patients with a history of mental illness or long-term psychiatric drugs (dementia, schizophrenia), chronic analgesic drug use history, alcoholism history and cognitive dysfunction;
3. any cerebrovascular accident occurred within 3 months, such as stroke, transient ischemic attack (TIA), etc.
4. Diabetic patients with severe diabetic complications (diabetic ketoacidosis, hyperosmolar coma, various infections, macrovascular disease, diabetic nephropathy);
5. Chronic hypoxia and carbon dioxide storage, such as chronic obstructive emphysema;
6. a long history of alcohol abuse;
7. Unable to cooperate to complete the test, the patient or family rejected the participant.

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients who met the inclusion and exclusion criteria for gastrointestinal surgery admitted to the Second Affiliated Hospital of Nanchang University.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-04-13 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
wave time-frequency analysis | one day before surgery, 7-10 days after surgery
  The characteristics of four kinds of brain wave α, β ,δ and θ were analyzed by professional EEG analysis software
P300 latency and peak changes | one day before surgery, 7-10 days after surgery
  The feature analysis of event-related potentials was carried out through professional EEG analysis software
EEG event-related potential accuracy and response time | one day before surgery, 7-10 days after surgery
  The accuracy of task EEG was analyzed statistically by using professional EEG analysis software
Incidence of postoperative short-term cognitive dysfunction | postoperative 1,3,6 months
  A telephone return visit was conducted on patients using the Revised Cognitive Function Telephone Questionnaire (TICS-M) at 1, 3, and 6 months after discharge.The total score was less than 28 points, which was considered as cognitive impairment.

SECONDARY OUTCOMES:
Systolic pressure | perioperative period
  "just entering the operating room", "immediately after intubation", "every 5 minutes after intubation until the patient leaves the operating room".
Diastolic pressure | perioperative period
  "just entering the operating room", "immediately after intubation", "every 5 minutes after intubation until the patient leaves the operating room".
Mean pressure | perioperative period
  "just entering the operating room", "immediately after intubation", "every 5 minutes after intubation until the patient leaves the operating room".
Heart rate | perioperative period
  "just entering the operating room", "immediately after intubation", "every 5 minutes after intubation until the patient leaves the operating room".
Maximum postoperative C-reactive protein (CRP) | Up to 1 month after surgery
  Only the highest CRP values detected in the normal course of gastrointestinal surgery are collected, and no additional blood sampling or interventions are performed
Minimum postoperative albumin | Up to 1 month after surgery
  Only the lowest albumin values detected in the normal course of gastrointestinal surgery are collected, and no additional blood sampling or interventions are performed
Postoperative pain | 1, 3, and 7 days after surgery
  The degree of postoperative pain was assessed using the Numerical Rating Scale (NRS). The pain level increased sequentially from 0-10
Complication | During the perioperative period, up to 1 month after surgery
  All the perioperative complications are recorded
Length of hospitalization | After the patient is discharged from the hospital, average 1 month
  The total number of days the patient spent at the hospital for the current consultation

CONTACTS AND LOCATIONS:
Overall Officials: Fuzhou Hua, Study Director — Second Affiliated Hospital of Nanchang University
Locations (1):
- the Second Affiliated Hospital of Nanchang University, Nanchang University, Jiangxi, NanChang, China